CLINICAL TRIAL: NCT07238010
Title: Understanding the Impacts and Experiences of Children Currently Experiencing Parental Imprisonment
Status: Not yet recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Elizabeth Paddock, Doctorate in Forensic Psychology Course Director, University of Nottingham
Other Study IDs: FMHS 160-0525
Record Dates: First submitted 2025-07-03; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Parental Imprisonment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Child participant: Participants who are above 16 years old with a parent in prison
  Interventions: Other: Parental Imprisonment
- Parent/Guardian: Non-offending parent or guardian of the child with a parent in prison
  Interventions: Other: Parental Imprisonment
- Professional: Professional working with the family or child with a parent in prison
  Interventions: Other: Parental Imprisonment

INTERVENTIONS:
Other: Parental Imprisonment — Participants who are currently experiencing parental imprisonment; either the child, non-offending guardian or parent, or professional. Child participants will be recruited whom already have a parent in prison. The professionals and non-offending parent/guardian of the child will be recruited.

SUMMARY:
This research aims to understand the impacts, experiences, and support needs of children who are aged 16 years and above, currently experiencing parental imprisonment from their own perspective, and from the perspective of their non-offending parent/caregiver/guardian and a professional. This research will adopt a case study design. Semi-structured interviews will be conducted with the child experiencing parental imprisonment, and the non-offending parent or caregiver. This research will also aim to recruit a professional working with the young person or family during parental imprisonment. This will be analysed interpretative phenomenological analysis.

DETAILED DESCRIPTION:
It is estimated that over 100,000 children in England and Wales are separated from their parents due to parental imprisonment, now recognised as an adverse childhood experience that can have multifaceted challenges for the families and children associated.

Separation from a parent under any circumstance can be experienced by a child as distressing and traumatic, however, researchers have likened the experience and impacts of parental imprisonment to losing a parent to death or divorce. Parental imprisonment is an ambiguous loss for a child, and is often characterised by the sudden loss of an attachment figure, however, this is coupled with stigmatisation and discrimination associated with offending. A considerable research base focusing on the non-offending partners has highlighted that the imprisonment of a loved one can result in experiences of disenfranchised grief, stigmatisation, and symptoms of trauma. It is possible that children may internalise the stigma attached to having a parent in prison, or the offence committed, which can result in low self-esteem, self-worth, and increased isolation, however, there remains scarce research focusing on children's experiences of parental separation by imprisonment, and how they make sense of this.

Utilising quantitative methods, research has found that parental imprisonment is associated with increased rates of mental health problems, major depression and attention disorders in comparison to the general population. Similarly, research has found that following parental imprisonment, children experienced depression, difficulties attending and concentration in school, chronic sleeplessness, loneliness, increased substance misuse, and financial challenges. In comparison to the general population, prisoners are also more likely to have experienced socioeconomic disadvantages, mental health problems, and marital difficulties, which are all found to be risk factors for mental health problems in children. Research supported this, suggesting that parental imprisonment has a disproportionate impact on children associated as a result of imprisonment magnifying existing social and economic disadvantages. It is therefore possible that pre-existing factors to parental imprisonment impact on child outcomes, and that parental imprisonment acts as a catalyst.

Despite a body of quantitative research attempting to understand the impacts of parental imprisonment on child outcomes, much is still unknown of a child's own experiences of parental imprisonment. An emerging evidence base has utilised qualitative methods with children, finding contrasting results. Children reported that parental imprisonment was a negative experience resulting in financial challenges, lack of support, and reduced academic opportunities, whilst others shared that parental imprisonment was a positive experience.

It is clear from the evidence base that children impacted by parental imprisonment are not a homogenous group, and research is required to understand the experiences of parental imprisonment on a child, within the context of individual risk and protective factors.

This research aims to understand the impacts, experiences, and support needs of children who are aged 16 years and above, currently experiencing parental imprisonment from their own perspective, and from the perspective of their non-offending parent/caregiver/guardian and a professional. This research will adopt a case study design. Semi-structured interviews will be conducted with the child experiencing parental imprisonment, and the non-offending parent or caregiver. This research will also aim to recruit a professional working with the young person or family during parental imprisonment. This will be analysed interpretative phenomenological analysis.

ELIGIBILITY:
Inclusion Criteria:

Adult Participant

* Is the parent/caregiver/guardian to a child (above 16 years old) currently experiencing parental imprisonment
* Participants are based in the UK (England, Wales, Scotland, or Northern Ireland), and have experienced parental imprisonment whilst in the UK.

Child Participant

* Child participants are above 16 years old at the time of data collection.
* Child participants are currently experiencing parental imprisonment.
* Participants are based in the UK (England, Wales, Scotland, or Northern Ireland), and have experienced parental imprisonment whilst in the UK.

Professional Participant

* Is a professional working with, or previously worked with the family or child impacted by parental imprisonment
* Has worked with the family or child impacted by parental imprisonment for at least one month.
* Participants are based in the UK (England, Wales, Scotland, or Northern Ireland), and have experienced parental imprisonment whilst in the UK.

Exclusion Criteria:

Adult Participant

* Are the parent of the child participant who was imprisoned.
* Not the current caregiver/guardian/parent to the child participant

Child Participant

* Child participants are the direct victim of their parental offence.
* The child participant is aware of their parent's offence and imprisonment.
* Below 16 years old at the time of data collection.

Professional Participant

• Professional participant is aware that the child's parent is in prison

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Impact of Parental Imprisonment Semi Structured Questionnaire | Through study completion, an average of 6 months
  What are the impacts and experiences of persons currently experiencing or supporting with parental imprisonment?

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Paddock, Dr, Study Chair — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beresford S, Loucks N, Raikes B. The health impact on children affected by parental imprisonment. BMJ Paediatr Open. 2020 Feb 10;4(1):e000275. doi: 10.1136/bmjpo-2018-000275. eCollection 2020. No abstract available. PMID 32154384

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT07238010/Prot_SAP_ICF_000.pdf